CLINICAL TRIAL: NCT06100536
Title: A Stand-alone Therapeutic Music-with-Movement Programme for People With Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Daphne Cheung, Associate Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HSEARS20211026009
Record Dates: First submitted 2023-09-27; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Cognitive Impairment
Keywords: Music-with-Movement; Music; Intervention; Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Music-with-movement intervention supported by the stand-alone music-with-movement system.
  Interventions: Behavioral: Music-with-movement

INTERVENTIONS:
Behavioral: Music-with-movement — The intervention group participants will receive 12 weekly music-with-movement interventions facilitated by trained staff in a community centre or a residential care home. The duration lasts 30 minutes to one hour. It can be carried out individually or with up to six persons in a group. The intervention will be supported by the standalone music-with-movement system.

SUMMARY:
The number of people living with cognitive impairment is increasing at an exponential rate. More than 100,000 older people are living with dementia in Hong Kong. Alarmingly, about 60% of long-term care residents or day-care centre users are living with dementia, nearly all of whom experience anxiety, depression, or other behavioural and psychological symptoms that place heavy demands on healthcare support and jeopardize their quality of life.

A standalone Music-with-Movement system is developed by integrating innovative and communication technology to facilitate the delivery of an evidence-based music-with-movement intervention. The technology employed are music library, 6-axis motion-sensing music instruments, wireless charging, and RFID.

This study aims to evaluate the changes in health outcomes (cognition, psychosocial well-being and perceived support) of older adults after receiving the service delivered by the trained staff using the standalone music-with-movement system.

DETAILED DESCRIPTION:
Methods:

1. Aims and objectives:

   1. to evaluate the feasibility of the system supporting staff from elderly care institutes in leading musical activities (i.e., recruitment, retention, and acceptability);
   2. to evaluate the engagement of the participants in the intervention; and
   3. to preliminarily examine the health conditions of older adults with cognitive impairment.
2. Methods:

   1. Design: Single-group pre-and-post-test design
   2. Participants: Older adults with cognitive impairment.
   3. Setting: Elderly care institutes, such as daycare centres, community centres, and/or nursing homes.
   4. Sample size: 750 participants.
   5. Outcomes: Recruitment rate, attrition rate, acceptability, any adverse events, engagement in the intervention, health outcomes (social support, frailty, health-related QoL, MoCA).
   6. Data analysis strategies:
   7. Ethical consideration: Approval has been obtained from the University (HSEARS20211026009)

ELIGIBILITY:
Inclusion Criteria:

* Older adults with cognitive impairment
* In a stable medical condition

Exclusion Criteria:

* With critical medical or psychiatric problems
* Those with uncorrectable hearing impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | through study completion, an average of 3 year
  Recruitment rate-defined as the proportion of eligible participants (following screening) who agreed to take part in the study (calculated as number of participants recruited (numerator)/number of eligible participants (denominator)).
  Reference: Easpaig, B. N. G., Zhai, J., Gray, R., Brown, E., & Bressington, D. (2022). Recruitment, attrition and intervention completion in clinical trials of psychosocial interventions involving people with early and emerging psychosis: a systematic review protocol. BMJ open, 12(9), e060863.
Attribution Rate | through study completion, an average of 3 year
  Attrition rate -defined as the proportion of participants at defined study points who discontinued the intervention or were lost to follow-up (calculated as number of participants that withdraw (numerator)/number of participants randomised (denominator)).
  Attrition rates will be calculated as three points: after randomisation, during the intervention and at final follow-up.
  Reference:
  Easpaig, B. N. G., Zhai, J., Gray, R., Brown, E., & Bressington, D. (2022). Recruitment, attrition and intervention completion in clinical trials of psychosocial interventions involving people with early and emerging psychosis: a systematic review protocol. BMJ open, 12(9), e060863.
Intervention completion rate | through study completion, an average of 3 year
  Intervention completion rate - defined as the proportion of participants who completed the allocated intervention (for at least 70% attendance). Calculated as number of participants allocated to the intervention that completed the minimum attendance (numerator)/number of participants allocated to treatment (denominator).

SECONDARY OUTCOMES:
Change in Multidimensional Scale of Perceived Social Support (MSPSS) Score | 6 months
  The Multidimensional Scale of Perceived Social Support ("MSPSS") is a 12-item instrument designed to measure an individual's perception of support from 3 sources: family, friends and a significant other (4 items for each subscale) (Zimet et al., 1988), rated on a 7-point Likert scale ranging from "1" Very Strongly Disagree to "7" Very Strongly Agree.
Change in Frail Scale | 6 months
  The scale is a short five-question assessment that can screen for frailty (Fatigue, Resistance, Ambulation, Illnesses, & Loss of Weight) (Abellan van Kan et al., 2008) . Scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status.
Change in Montreal Cognitive Assessment 5-minute (MoCA) | 6 months
  The 5-minute "Mini MoCA" is an abbreviated version of MoCA, composed of the tasks proven most sensitive to mild cognitive impairment. The MoCA 5-min protocol in Cantonese version was validated to be reliable cognitive screening tools (Wong et al., 2015).
Change in Health-related Quality of Life (EQ-5D-3L) | 6 months
  The EQ-5D-3L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression (EuroQol Group). Each dimension has 3 levels: no problems, some problems, and extreme problems. The total score of five items can describe the patient's health state. Also, the participants are asked to self-rating their health state on a vertical visual analogue scale (0 = the worst health state to 100 = the best health state) to reflect their own judgement.
Change in Neuropsychiatric Symptoms - Informant-based | 6 months
  This is an informant-based instrument that measures the presence and severity of 12 neuropsychiatric symptoms in older adults with cognitive impairment and their associated distress over the previous month (Kaufer et al., 2000).
Engagement during the intervention | 3 months
  Trained research assistant will observe the participants' engagement level during the intervention measured with Non-pharmacological Therapy Experience Scale (overall score ranges 0 - 30). Higher score means better engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Sze Ki Cheung, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided